CLINICAL TRIAL: NCT00734812
Title: LSH vs. TLH, A Randomized Single Blind Trial
Brief Title: Laparoscopic Supracervical Hysterectomy Versus Total Laparoscopic Hysterectomy
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was withdrawn prior to any enrollment.
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Jon I. Einarsson, Chief, Division of Minimally Invasive Gynecology, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2007-P-002591/1
Record Dates: First submitted 2008-08-12; First posted 2008-08-14 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Gynecologic Diseases
Keywords: Hysterectomy; Laparoscopic
MeSH Terms: conditions — Genital Diseases, Female

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Laparoscopic supracervical hysterectomy (LSH)
  Interventions: Procedure: Laparoscopic supracervical hysterectomy
- 2 (Active Comparator): Total Laparoscopic Hysterectomy (TLH)
  Interventions: Procedure: Total laparoscopic hysterectomy

INTERVENTIONS:
Procedure: Laparoscopic supracervical hysterectomy — Patients will be randomized to LSH (retaining the cervix) and TLH (cervix removal)
  Arms: 1
Procedure: Total laparoscopic hysterectomy — Patients will be randomized to either removal or retention of cervix
  Arms: 2

SUMMARY:
The purpose of this research study is to evaluate whether there is any difference in recovery time and return to normal activities following a laparoscopic supracervical hysterectomy (LSH) compared with total laparoscopic hysterectomy (TLH). Both types of hysterectomies are commonly performed at our institution.

Patients will be assigned by chance (like a coin toss) to have either a LSH or a TLH. Preoperatively, participants will complete a quality of life questionnaire (SF-36), a sexual function questionnaire (FSFI)and a 3 question questionnaire about urinary function (3IQ).

Following surgery participants will be asked to keep a diary of pain symptoms and use of narcotics. The diary will be filled out daily until patients have resumed normal activities from prior to the surgery. The SF-36 will be completed again 6 weeks following the original surgery.

6 months following surgery participants will receive a copy of the SF-36 and the FSFI in the mail. They will also be asked questions about urinary symptoms and persistent vaginal bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for laparoscopic hysterectomy for benign indications

Exclusion Criteria:

* Malignancy of the uterus, cervix or adnexa
* pre-malignant changes of the uterus, cervix or adnexa
* history of severe cervical dysplasia (CIN II or above)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-05; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Return to normal activities | 3-6 weeks after surgery

SECONDARY OUTCOMES:
Sexual function | 6 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jon I. Einarsson, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States